CLINICAL TRIAL: NCT03743103
Title: A Randomized, Exploratory, Open-label, Phase IV, Blinded Endpoint, Multicenter and Prospective Study to Evaluate the Effect of the Addition of Esmolol on the Current Therapeutic Regimen Used for the Treatment of Hemorrhagic Stroke
Brief Title: Esmolol for the Treatment of Hypertension After Intracerebral Hemorrhage Study (ETHICHS)
Acronym: ETHICHS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollement
Sponsor: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRT088
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Hemorrhagic Stroke
MeSH Terms: conditions — Hemorrhagic Stroke | interventions — esmolol; Nitroprusside

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brevibloc, 10 Mg/mL Intravenous Solution (Experimental): 10 mL/h every 5 minutes until reaching the pressure target
  Interventions: Drug: Brevibloc, 10 Mg/mL Intravenous Solution; Drug: Nitroprusside, Sodium
- Nitroprusside, Sodium (Active Comparator): 0.5 mcg / kg / min every 3 minutes until reaching the pressure target
  Interventions: Drug: Nitroprusside, Sodium

INTERVENTIONS:
Drug: Brevibloc, 10 Mg/mL Intravenous Solution — 10 mL/h every 5 minutes until reaching the pressure target
  Other Names: Brevibloc
  Arms: Brevibloc, 10 Mg/mL Intravenous Solution
Drug: Nitroprusside, Sodium — 0.5 ug/kg/min every 3 minutes until reaching the pressure target
  Other Names: Nitroprus

SUMMARY:
Because of its pharmacokinetic characteristics, such as short half-life and its safety profile, esmolol hydrochloride is a beta blocker suitable for venous use in the form of continuous infusion. Strategies that improve the blood pressure control of patients with hemorrhagic stroke during the first hours of hospitalization are determinant in controlling the hematoma expansion and determining factor in its prognosis. This study was designed with the objective of evaluating the beneficial effects of combining esmolol hydrochloride with sodium nitroprusside for the blood pressure control of participants with hemorrhagic stroke.

DETAILED DESCRIPTION:
Participants with parenchymal intracranial hemorrhage (diagnosis confirmed by computed tomography or magnetic resonance imaging), and:

* with systolic pressure > 150 mmHg,
* not contraindicated for treatment with beta-blockers,
* who can start the drug treatment within 6 hours of the stroke,
* having a target of ≤ 140 mmHg of systolic pressure within 1 hour after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signature of the TCLE by participant or companion.
2. Spontaneous intracerebral hemorrhage confirmed by computed tomography or magnetic resonance imaging and fit to be included in the study and initiate therapy with study medications within 6 hours after the event.
3. Intracerebral hemorrhage (volume < 30 cm3).
4. No immediate surgical indication.
5. Both sexes, aged above 18 years.
6. Systolic blood pressure (> 150 mmHg and < 220 mmHg) measured on two occasions with a minimum difference of 2 minutes.

Exclusion Criteria:

1. Cerebral hemorrhage secondary to structural lesions in the brain, vascular malformations, coagulopathies or traumatic brain injury, if known at the time of randomization.
2. Participant in deep coma, defined by the Glasgow Coma Scale score of 3 to 5.
3. Uncontrolled asthmatic or COPD participants, if known at the time of randomization.
4. Participants with Grade IV Heart Failure, defined as heart rate < 50 beats per minute.
5. Previous hemorrhagic stroke, if known at the time of randomization
6. Participants with Cerebral Vascular Stroke.
7. Participants who have presented previous ischemic cerebrovascular accident, if known at the time of randomization.
8. Chronic diseases with life expectancy less than 3 months.
9. Score ≥ 4 on the ICH score at the time of recruitment.
10. In use of anticoagulants in the last 48 hours, if known at the time of randomization.
11. Patients with contraindication to any of the study medications.
12. Intubation Orotraqueal on arrival at the service.
13. Pheochromocytoma, if known at the time of randomization.
14. Patients with hyperthyroidism, if known at the time of randomization.
15. Known pregnancy or breastfeeding . At the discretion of the investigator, an examination for confirmation may be requested.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
To evaluate comparatively the drug test and the comparator drug | 7 days
  Variation of systolic and diastolic pressure during the time of use of the investigational products measured by ABPM (outpatient blood pressure monitoring).

SECONDARY OUTCOMES:
To compare the percentage of participants | in the first hour of treatment between the groups.
  To compare the percentage of participants with controlled systolic pressure (goal ≤ 140 mmHg)
Rankin Scale | in 90 ± 4 days
  To compare the ranks of the modified Rankin Scale (Applied by blind-investigator) between groups.
NIH Stroke Scale (NIHSS) and Glasgow Coma Scale | from admission to discharge or 7th day
  Compare the variation in scores on the NIH Stroke Scale (NIHSS) and Glasgow Coma Scale (whichever comes first) between groups.
MOCA scale | in 90 ± 4 days
  To compare the cognitive performance assessed between the groups.
Hematoma volume expansion and perihematoma volume of cerebral edema | 24 ± 4 hours
  To compare the percentages of between admission tomography and control tomography after the end of infusion of investigational products
Severe hypotensive events with clinical consequences | in 90 ± 4 days
  To compare the frequency of severe hypotensive events with clinical consequencesrequiring corrective therapy with vasopressors during the use of investigational products between groups.
Adverse events related with investigational product | in 90 ± 4 days
  To compare the frequency and intensity of adverse events related to the use of research products between groups.
Severe cardiovascular events | in 90 ± 4 days
  Compare the frequency of severe cardiovascular events (acute myocardial infarction, cardiac arrest, arrhythmias, or the development of severe congestive heart failure) or major neurological complications (eg need for neurosurgery, intraventricular bypass placement, cerebral infarction, convulsive seizures, intoxication, neurological toxicity) within the first 90 days of follow-up between groups.
Bradycardia | in 90 ± 4 days
  Compare the frequency and duration of major bradycardia (<50 beats per minute) between groups.
QT interval variability | during the infusion period
  Compare the QT interval variability measured by Holter during the infusion period of the investigational products between the groups
Frequency of changes in the ECO | in the first 72 ± 4 hours and the return after 90 ± 3 days
  Compare the frequency of changes in the Echocardiogram (Differences observed between the examination performed in the first 72 ± 4 hours and the return after 90 ± 3 days) between the groups.
Frequency of changes in the level of BNP | at baseline times, 24 ± 4 and 72 ± 4 hours
  To compare the frequency of changes in the level of B-type natriuretic peptide (BNP) measured at baseline times, 24 ± 4 and 72 ± 4 hours between groups.
Frequency of changes in baseline cardiac troponin levels | 24 ± 4 and 72 ± 4 hours
  To compare the frequency of changes in baseline cardiac troponin levels, 24 ± 4 and 72 ± 4 hours
Frequency of intra-cranial hypertension | 7 days
  To compare the frequency of intra-cranial hypertension diagnosed by measuring the diameter of the optic nerve sheath by transorbital ultrasound daily for 7 days or high, whichever occurs first between the groups.

CONTACTS AND LOCATIONS:
Locations (7):
- Brazil (7):
  - Hospital Geral de Fortaleza, Fortaleza, Ceará
  - Hospital São Rafael, Salvador, Estado de Bahia
  - Hospital Madre Teresa, Belo Horizonte, Minas Gerais
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas da Faculdade de Medicina de Botucatu, Botucatu, São Paulo
  - Hospital das Clínicas de Riberião Preto, Ribeirão Preto, São Paulo
  - Universidade Federal de São Paulo, São Paulo